CLINICAL TRIAL: NCT04331678
Title: Evaluation of a Mobile App to Promote Social Support for Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Cancer Center (Other)
Collaborators: Pfizer (Industry); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-002b
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Chemotherapy Effect

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants will be complete survey at enrollment and then again in 3 months.
- Active (Active Comparator): Participants in the App group will receive usual care and complete survey at enrollment and then again in 3 months.
  In addition, they will be asked to download the study app to their mobile device and use it at least once per week during the 3-month study period.
  Interventions: Behavioral: Comparator App

INTERVENTIONS:
Behavioral: Comparator App — Participants will download and agree to use the study app at least once per week during the 3-month intervention period.
  The app allows participants to invite a network of friends and family to provide emotional and logistical support during their treatment.
  Arms: Active

SUMMARY:
Our study will evaluate patient and caregiver use of a new mobile application (app) to support patients undergoing chemotherapy treatment for cancer.

DETAILED DESCRIPTION:
The app is designed to be used by the patient and members of their support network. It provides wide-ranging functionality, including: reminders for appointments and tasks, the ability to track health measures (fitness, emotion, pain, sleep), archive health related documents, maintain notes and recordings from visits, social networking functions to connect with family and friends to coordinate support activities and share news, and educational resources. We will randomize 230 patients initiating chemotherapy cancer treatment and up to one caregiver to the App group (asked to use the app once or more per week) or the Usual Care group, and evaluate the 3-month efficacy of app use on key outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Patients must have a confirmed diagnosis of cancer and be prior to or within one month of initiating chemotherapy or immunotherapy
* Have a valid email address
* Have a smart mobile device (Android or iOS) with a data plan
* Willing to download and use the study app

Exclusion Criteria:

* Unable to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2021-10-24 (Actual)

PRIMARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy-General (FACT-G) Score | Baseline, Three months
  a. Investigators will measure the relative changes in functional status of cancer patients using the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire. FACT-G is a 27-item questionnaire asking participants to report the four primary QoL domains, including physical, social/family, emotional and functional well-being on a 5-point Likert scale where 0 = Not at all to 4 = Very much with higher scores representing better general QoL.
Change in Short-Form Health Survey (SF-12) | Baseline, Three months
  a. Investigators will measure differences in quality of life between the two study arms with the SF-12 instrument. The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. SF-12 is a standardized self-report questionnaire that assesses mental and physical functioning. The SF-12 consists of 12 items with a Likert-type response format that measures quality of life with a Physical Component Summary (PCS) and Mental Component Summary (MCS). Subscales associated with the PCS include physical functioning, role limitations due to physical problems, bodily pain, and general health perceptions. Subscales associated with the MCS include vitality (energy and fatigue), social functioning, role limitations due to emotional problems, and mental health. A scoring algorithm is used to generate a total score for each component ranging from 0 to 100. Low values represent a poor health state while high values represent a good health state.

SECONDARY OUTCOMES:
Caregiver's Burden | Baseline, Three months
  Changes in the caregiver's burden assessed using the 10-item Caregiver Quality of Life - Cancer Scale (CQOLC) Burden Subscale, where higher scores indicate greater burden.
Caregiver's Disruptiveness | Baseline, Three months
  Changes in the caregiver's disruptiveness of daily life will be assessed using the 7-item CQOLC Disruptiveness Subscale, where scores are calculated as described for burden, and higher scores indicate greater disruptiveness.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - West Cancer Center, Southaven, Mississippi
  - West Cancer Center, Germantown, Tennessee
  - West Cancer Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graetz I, Hu X, Curry AN, Robles A, Vidal GA, Schwartzberg LS. Mobile application to support oncology patients during treatment on patient outcomes: Evidence from a randomized controlled trial. Cancer Med. 2023 Mar;12(5):6190-6199. doi: 10.1002/cam4.5351. Epub 2022 Oct 18. PMID 36258654